CLINICAL TRIAL: NCT04861636
Title: Enhancing Emotion Regulation to Support Weight Control Efforts in Adolescents With Overweight and Obesity
Brief Title: Teen Weight Control
Acronym: HealthTRAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Rhode Island Hospital (Other); University of Oregon (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK12455101
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Obesity; Weight Loss
MeSH Terms: conditions — Pediatric Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Both the standard behavioral weight control (SBWC) and HealthTRAC interventions include 4 months of intensive treatment, followed by monthly maintenance sessions for a 12-month program. SBWC includes attention to diet and activity coupled with behavioral modification strategies. HealthTRAC integrates these key constructs with an emotion regulation intervention with documented efficacy in teens.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthTRAC (Experimental): Both the standard behavioral weight control (SBWC) and HealthTRAC interventions include 4 months of intensive treatment, followed by monthly maintenance sessions for a 12-month program. SBWC includes attention to diet and activity coupled with behavioral modification strategies. HealthTRAC integrates these key constructs with an emotion regulation intervention with documented efficacy in teens.
  Interventions: Behavioral: HealthTRAC
- Standard Behavioral Weight Control (SBWC) (Active Comparator): 4 months of intensive treatment focused on attention to diet and activity coupled with behavioral modification strategies, which is then followed by monthly maintenance sessions for a 12-month program.
  Interventions: Behavioral: SBWC

INTERVENTIONS:
Behavioral: HealthTRAC — Behavioral weight management intervention targeting emotion regulation skill building. Intervention components will be delivered in 27.5 hours of direct contact time across 12 months. All adolescents will be assessed prior to randomization (baseline), immediately following the intervention (4 months), upon completion of maintenance sessions (12 months) and 18 months after the start of intervention.
  Arms: HealthTRAC
Behavioral: SBWC — Behavioral intervention focused on behavioral weight control. Intervention components will be delivered in 27.5 hours of direct contact time across 12 months. All adolescents will be assessed prior to randomization (baseline), immediately following the intervention (4 months), upon completion of maintenance sessions (12 months) and 18 months after the start of intervention.
  Arms: Standard Behavioral Weight Control (SBWC)

SUMMARY:
The prevalence of obesity in adolescents is remarkably high, with 38.7% of youth 12-15 years of age and 41.5% of 16-19 year olds meeting criteria for overweight or obesity. Behavioral weight control interventions for adolescents have had limited impact on this field and there is considerably more that needs to be done. Notably, adolescents who have difficulty managing their feelings have been found to consume higher caloric foods and report greater amounts of sedentary time. Poor emotion management among adolescents has also been associated with more rapid weight gain and higher BMI. Data from adolescents with overweight/obesity attending our outpatient weight management program (N=124) indicate that 82% of these youth report emotion regulation scores that are comparable to youth with significant mental health problems. Despite documented relationships between adolescent weight control and emotion regulation, no proven adolescent weight management programs targeting emotion regulation exist. To fill this gap, our laboratory developed and piloted an adolescent weight control intervention (HealthTRAC) that combines two previously tested effective interventions, one targeting emotion regulation skill building, the other focused on behavioral weight control. Findings from our small pilot trial are promising and indicate that the newly created HealthTRAC intervention is acceptable to parents and teens, easy to deliver, and leads to modest weight loss and improved emotion management skills compared to a standard behavioral weight control (SBWC) program. These data suggest that emotion regulation is related to weight management and may assist adolescents with overweight/obesity who are seeking to lose weight. The current multi-site study builds on this previous work and will examine the impact of the developed HealthTRAC intervention on improving emotion regulation skills and reducing adolescent BMI in a larger sample with longer term follow-up (18 months after starting the intervention). Adolescents will receive 27.5 hours of intervention time over a 12- month period. We expect that adolescents enrolled in the HealthTRAC intervention will show greater reduction in BMI over the 12-month program and will sustain these losses up to 18 months after starting the intervention compared to teens enrolled in SBWC. The information learned from this project will help us better understand how helping adolescents manage their emotions can improve weight loss outcomes.

DETAILED DESCRIPTION:
Participants will be assigned to one of two treatment conditions (HealthTRAC or Standard Behavioral Weight Control) using urn randomization procedure. Participants assigned to either condition will receive a 12-month weight control intervention that includes 12 weekly sessions and 2 bi-weekly sessions (14 primary sessions delivered over 4-months), followed by 8 months of maintenance sessions. Both conditions will also include parents at sessions 1, 7, and 14, and maintenance sessions at 6-8-,10-, and 12 months.

Both interventions will be delivered using a group-based treatment model. We selected a control condition that offers a more rigorous test of the program than a treatment as usual condition, commonly included in efficacy trials. Few studies have examined the combined impact of targeting emotion regulation skills and standard behavioral weight control strategies. Given the literature documenting the relationship between emotion regulation and weight-related behaviors, and the evidence from adult weight management studies, targeting this construct in adolescent populations may facilitate improved weight management outcomes via a reduction in emotional eating and sedentary time and improvement in overall diet quality.

The timing of study assessments immediately following intervention and at 12 months are justified by improvements in primary weight status outcomes observed in the treatment development study that was the immediate precursor of the proposed trial. Our previous work delivering adolescents weight control interventions supports our ability to retain participants through this study period. We have included an 18-month follow-up to examine sustainability of intervention effects. Few weight control interventions with adolescents include outcomes out to 18 months, and those that do, often have low rates of retention. Following established protocols, we anticipate approximately 80% retention at 18-month follow-up.

Participants will be enrolled into the efficacy trial continuously between Year 1, Month 6 and Year 4, Month 37. Consistent with the HealthTRAC pilot trial, we will recruit participants from primary care clinics and subspecialty clinics affiliated with children's hospitals, as well as through community advertisements. The majority of adolescent referrals to the treatment development study came from pediatric health care clinics at Hasbro Children's Hospital in Providence, RI (90%), with local advertisements accounting for the remainder. We anticipate that health care clinics will serve as a primary source for recruitment for the current trial. We will use parallel procedures to enroll participants in Providence, RI and Portland, OR. The PIs will work with representative staff from Hasbro Children's Hospital (RI) and Doernbecher Children's Hospital (OR) to distribute Consent to Contact forms, which can be completed by interested families. Families recruited in these settings will receive follow-up calls, emails, or texts (based on preference) to further determine initial eligibility and schedule consent/assents. Study brochures and advertisements will also be sent to adolescents who receive care within these various settings via direct home mailings. In addition to these successful approaches from the HealthTRAC pilot trial, we will also advertise through Facebook ads directed at parents. This strategy has been very effective in recent enrollment of adolescents to a behavioral weight control trial.

Initial evaluations will be conducted at the Weight Control and Diabetes Research Center or the University of Oregon Portland campus. Parents will undergo a brief interview and parents and adolescents will complete questionnaire measures. Adolescents will also complete computerized emotion regulation tasks. Parent questionnaires will focus on socio-demographic variables, the teen's dieting and medical history, any psychiatric history and treatment and emotion regulation abilities. Adolescent questionnaires will focus on emotion regulation abilities, mental health symptoms, and emotional eating. The first of the 24-hour dietary recalls will also be conducted during this visit, and adolescents will be provided instruction regarding completing 7-day accelerometry. Adolescent height and weight will be obtained at the end of the evaluation. Participants will be asked to return accelerometers after one week of wear or at the first intervention session, depending on the timing. Adolescents and parents will be informed of randomization condition at the first intervention session.

Most of the baseline battery will be re-administered post treatment, 12-, and 18-month follow-ups by an assessor masked to the baseline results and treatment assignment. In order to increase convenience, every effort will be made to conduct follow-up evaluations at the conclusion of intervention sessions or at times convenient for families (18-month assessment). This approach has been effective in both our previous weight control and adolescent emotion regulation trials. Assessments may be conducted on weekend mornings to avoid disruption to school attendance.

For the adolescent group interventions, the adherence measure developed in the pilot trial for HealthTRAC will be used. All efficacy trial sessions will be videotaped. We have chosen to videotape sessions in order to capture both verbal and nonverbal aspects of participant ad interventionist interactions, especially relevant for the emotion regulation skill building components of the HealthTRAC intervention.

The HealthTRAC intervention was tested in an open trial with youth 13 - 17 years of age and in a recently completed treatment development study that included a small randomized controlled trial with adolescents (R21 DK108164). The HealthTRAC intervention combined two efficacious interventions that separately targeted adolescent weight management (SBWC: R01HL6513201; R01DK062916) and adolescent emotion regulation skill building (TRAC; R01 NR011906). We will use procedures established in our previous work to ensure that the intervention is administered in a standardized manner across groups.

The goals of the HealthTRAC intervention are to facilitate improved emotion regulation abilities with the goal of promoting healthy pediatric weight management. This will be achieved in accordance with goals established by the American Academy of Pediatrics (AAP) guidelines that support modest weight loss for youth with BMI greater than or equal to the 95th percentile. These guidelines serve as the principles on which both interventions are based. Reductions in weight status are supported by recommended calorie reductions established in pediatric samples and are as follows:

150 lbs. or less 1200 - 1400 calories 151-249 lbs. 1400 - 1600 calories 250 lbs. and more 1600 - 1800 calories

Activity goals prescribed through the intervention are commensurate with current activity guidelines for youth and include gradually increasing moderate-to-vigorous physical activity to 60 minutes daily and decreasing sedentary behavior to no more than two hours per day.

Specific content included over the course of the intensive weekly curriculum include: (1) orientation to the program and self-monitoring, (2) energy balance and nutrition goals, (3) stimulus control, (4) physical activity and sedentary behavior, (5) diet quality, (6) ding it on your own and self-motivation, (7) behavior chains and problem solving, (8) eating outside the home, (9) timing of eating occasions and coping with cravings, (10) developing and maintaining a healthy body image, (11) managing holidays, vacation, and special occasions, (12) cultural and social influences, (13) relapse prevention, and (14) review and transition to monthly sessions.

Content covered during the course of the maintenance sessions include managing daily challenges, moods and foods, managing peer interactions, maintaining motivation, tricks and tips, myth busters, and undoing small weight gains.

Lesson Format: Each session will last 75 minutes. The first 15 minutes will be devoted to adolescent weigh-ins and review of self-monitoring records. The remaining 60 minutes is focused on the specific weekly content, with 10 minutes at the end of each session dedicated to setting goals and problem solving relevant to the week;s lesson. While these are approximate times, the allocation clearly indicates the emphasis placed on problem-solving and overcoming challenges throughout the curriculum.

We will also employ our previously used strategy of awarding points for gradual weight loss, achievement of self- selected dietary or physical activity goals, and submission of weekly food diaries, which was also endorsed in adolescent interviews, to support retention of participants through the maintenance phase. Incentivizing weight loss behaviors and weight loss has been demonstrated to be an effective strategy in previous trials and was therefore implemented within the pilot trial and will be retained for the current proposal.

HealthTRAC Specific Format: Within emotion regulation training intervention emotion regulation skills are incorporated into the weigh-in. Facilitators prompt each participant to identify bodily cues associated with emotions prior to stepping on the scale and review potential emotions that could have interfered with previously set weekly goal.

Emotion regulation training skills are taught across the first 7 sessions of the program, and specific activities linking emotion regulation to dietary behaviors are utilized across all remaining sessions across specific mood induction tasks.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants must:

1. be between 13 and 17 years of age
2. have BMI greater than or equal to the 95th percentile for age and sex
3. have a parent or guardian available to participate in the study
4. speak English due to the group format of the intervention
5. agree to study participation, measures, and randomization
6. be available for long-term follow-up.

EXCLUSION CRITERIA:

Adolescents will be excluded from study participation if they:

1. have absolute BMI greater than 50
2. are currently involved with another weight loss program
3. have a medical condition that would interfere with the prescribed dietary plan or participation in physical activity
4. have a developmental delay such that the intervention materials will not be appropriate
5. report engaging in extreme/unhealthy weight control behaviors including self-induced vomiting, laxative or diuretic use, or report a history of eating disorder, and/or are actively psychotic or suicidal at the time of screening.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in BMI from baseline to 12 months post-intervention | baseline and 12 months after randomization
  Weight (kilograms) and height (meters^2) will be used to calculate body mass index (BMI; kg/m^2)

SECONDARY OUTCOMES:
Examine the impact of HealthTRAC relative to SBWC on emotion regulation | baseline and 4-, 12-, 18- months after randomization
  Completed by adolescents, DERS assesses six domains of emotion regulation on a five-point Likert scale, three of which are germane to our construct (Strategies, Impulses, and Goals). The Emotion Regulation Behaviors Scale (ERBS) assesses the use of the specific emotion regulation strategies taught in our interventions. Completed by both parents and adolescents, the Affect Dysregulation Scale (ADS) assesses the frequency of adolescents' difficulties with affect regulation. Completed by parents, the Emotion Regulation Checklist (ERC) is a measure of adolescents' emotion regulation from the perspective of the parent/caregiver. Two subscales are generated (Lability/Negativity and Emotion Regulation). Completed by adolescents, the Behavioral Indicator of Resiliency to Distress (BIRD) is a computerized distress tolerance task. This measure generates a score of total time that adolescents persist on a frustrating computerized task, which has been linked to emotion regulation abilities.
Examine the impact of HealthTRAC relative to SBWC on emotional eating | baseline and 4-, 12-, 18- months after randomization
  The Emotional Eating Scale is a 25-item self- report measure used to assess the propensity to cope with emotions by eating. Subscales include: Eating in response to anxiety, anger, and frustration (AAF), depressive symptoms (DEP), and feeling unsettled (UNS). One additional item assesses eating in response to positive affect ("happy"). For a more nuanced assessment, we will administer a 5-item assessment via secure Qualtrics link for 7 days during each assessment period. Teens will be asked to reflect on whether they experienced eating in response to any of five emotions during the course of the day. (i.e., sadness, anxiety or worry, boredom, happiness, or frustration).
Examine the impact of HealthTRAC relative to SBWC on dietary intake | baseline and 4-, 12-, 18- months after randomization
  Dietary Intake will be measured via three, non- consecutive 24-hour diet recalls. Each recall will be collected via a software program that employs a variation of the USDA's validated Multiple Pass Method to collect detailed information on each food and beverage consumed at each eating occasion over the previous 24-hour period. Data will be used to calculate Healthy Eating Index.
Examine the impact of HealthTRAC relative to SBWC on physical activity and sedentary behavior | baseline and 4-, 12-, 18- months after randomization
  Physical Activity and Sedentary Behavior will be assessed with accelerometer (ActiGraph, LLC, Pensacola FL) for a 1-week period at each of the primary assessment points.
Examine the impact of HealthTRAC relative to SBWC on screen time | baseline and 4-, 12-, 18- months after randomization
  Screen time will be assessed using 7 items derived from The Common Sense Census: Media Use by Tweens and Teens (2019). Items assess both type and amount of screen time during the previous day. This will be administered at the end of each 24-hour dietary recall interview.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Jelalian, PhD, Principal Investigator — Elissa_Jelalian@brown.edu
Locations (3):
- United States (3):
  - University of Oregon, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04861636/ICF_000.pdf